CLINICAL TRIAL: NCT04574492
Title: Canadian Real-life Post-marketing Observational Study Assessing the Effectiveness of Upadacitinib for Treating Rheumatoid Arthritis (CLOSEUP)
Brief Title: A Study of Oral Upadacitinib Tablets to Assess the Change in Disease Symptoms in Adult Canadian Participants With Moderate to Severe Rheumatoid Arthritis
Acronym: CLOSEUP
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-096
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis; Upadacitinib; RINVOQ
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants receiving Upadacitinib: Participants receiving Upadacitinib for moderate to severe rheumatoid arthritis (RA).

SUMMARY:
Rheumatoid Arthritis (RA) is an inflammatory disease of the joints causing pain, stiffness, swelling and loss of joint function. This study will assess how effective Upadacitinib is in changing the disease symptoms in Canadian participants with RA.

Upadacitinib is a drug approved for the treatment of moderately to severely active rheumatoid arthritis. Adult Canadian participants with moderate to severe RA who have been prescribed upadacitinib by their physicians will be enrolled. Approximately, 390 participants will be enrolled this study, in multiple sites within Canada.

Participants will receive Upadacitinib as prescribed by the physician and will be followed for approximately 24 months.

There will be no additional burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic and will be asked to provide additional information by questionnaire at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe Rheumatoid Arthritis (RA) according to the investigator.
* Decision to initiate UPA treatment by investigator according to the local product label independent of the participant's participation in the study.
* Has been previously treated with Conventional Synthetic Disease-Modifying Antirheumatic Drugs (csDMARDs) and corresponds to one of the following subgroups:

  * Has not been previously exposed to any Biologic Disease-Modifying Antirheumatic Drugs (bDMARD) or Targeted Synthetic Disease-Modifying Antirheumatic Drugs (tsDMARD).
  * Has not been previously exposed to tsDMARD and has been previously exposed to <= 2 bDMARDs.
  * Has been previously treated with one tsDMARD and <=1 bDMARD prior to treatment with that tsDMARD.

Exclusion Criteria:

* Presence of any condition that, in the opinion of the treating physician, prohibits the participant from participating in the study or obscures the assessment of the treatment of RA.
* Diagnosis of rheumatic disease other than RA.
* Diagnosis of juvenile RA.
* Currently participating in an investigational clinical trial.
* Has prior exposure to a bDMARD after exposure to a tsDMARD.
* Has prior exposure to tsDMARD in an investigational clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants receiving Upadacitinib according to the product prescribing information, for moderate to severe active Rheumatoid Arthritis (RA).
Sampling Method: Non-Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieve Clinical Remission | At Month 6
  Clinical remission is defined as Disease Activity Score at 28 joints (DAS28) C-reactive Protein (CRP)<2.6.

SECONDARY OUTCOMES:
Change in Pain Using Visual Analogue Scale (VAS) | Baseline (Month 0) Through Month 24
  Pain is defined using VAS, where a higher score indicates worse pain.
Duration of Morning Stiffness | Baseline (Month 0) Through Month 24
  Duration of morning joint stiffness is defined using VAS, where a higher score indicates worse joint stiffness.
Severity of Morning Stiffness | Baseline (Month 0) Through Month 24
  Severity of morning joint stiffness is defined using VAS, where a higher score indicates worse joint stiffness.
Change in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | Baseline (Month 0) Through Month 24
  The FACIT Fatigue Scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four-point Likert scale (0 = not at all fatigued to 4 = very much fatigued).
Percentage of Participants Achieving Clinical Remission | Baseline (Month 0) Through Month 24
  Clinical Remission is defined as DAS28-CRP<2.6, Simplified Disease Activity Index (SDAI) ≤3.3, Clinical Disease Activity Index (CDAI) ≤2.8, American College of Rheumatology (ACR)-European League Against Rheumatism (EULAR) Boolean remission.
Percentage of Participants Achieving Low Disease Activity (LDA) | Baseline (Month 0) Through Month 24
  LDA is defined as DAS28-CRP<3.2, SDAI ≤11, CDAI ≤10.
Earliest Date When a Response to Treatment is Known to Have Occurred | Baseline (Month 0) Through Month 24
  Earliest date when a response to treatment is known to have occurred.
Earliest Date When Their RA is Known to have Returned (In those Participants who Achieve a Response to Treatment) | Through Month 24
  Earliest date when their RA is known to have returned (In those participants who achieve a response to treatment).
Change in DAS28-CRP Score | Baseline (Month 0) Through Month 24
  The DAS28-CRP used to evaluate disease activity in participants with RA, where worsening RA activity is defined by a higher score.
Change in CDAI Score | Baseline (Month 0) Through Month 24
  The CDAI is used to evaluate disease activity in participants with RA , where worsening RA activity is defined by a higher score.
Change in Tender Joint Count | Baseline (Month 0) Through Month 24
  Change in Tender Joint Count.
Change in Swollen Joint Count | Baseline (Month 0) Through Month 24
  Change in Swollen Joint Count.
Change in Physical Function (HAQ-DI) Score | Baseline (Month 0) Through Month 24
  The HAQ DI is a questionnaire that determines physical function.
Change in Patient Assessment of Global Disease Activity (PtGA) | Baseline (Month 0) Through Month 24
  The PtGA is a outcome instrument to assess the participant's assessment of disease severity.
Change in Physician Assessment of Global Disease Activity (PGA) | Baseline (Month 0) Through Month 24
  The PGA is a outcome instrument to assess the participant's assessment of disease severity.
Percentage of Participants Who Discontinue Upadacitinib | Through Month 24
  Percentage of participants who discontinue Upadacitinib.
Time of Discontinuation from Upadacitinib Initiation Date | Through Month 24
  Time of discontinuation from Upadacitinib initiation date.
Reasons for Upadacitinib Treatment Discontinuation | Through Month 24
  Reasons for Upadacitinib treatment discontinuation.
Immediate Change in RA Medications Following Discontinuation of Upadacitinib | Through Month 24
  Immediate change in RA medications following discontinuation of Upadacitinib.
Percentage of Participants Who Achieve Sustained Remission Following Discontinuation of Upadacitinib | Through Month 24
  Clinical remission is defined as DAS28 and CRP<2.6.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (39):
- Canada (39):
  - Rheumatology Research Associates /ID# 224534, Edmonton, Alberta
  - Saurash Reddy Professional Corporation /ID# 225288, Edmonton, Alberta
  - Fraser Clinical Trials Inc /ID# 225200, New Westminster, British Columbia
  - Dr. Jonathan D. Chan Inc. /ID# 222976, Vancouver, British Columbia
  - Dr. Milton F. Baker Inc. /ID# 224555, Victoria, British Columbia
  - Manitoba Clinic /ID# 223288, Winnipeg, Manitoba
  - Eastern Regional Health Authority /ID# 223911, St. John's, Newfoundland and Labrador
  - Nexus Clinical Research /ID# 225896, St. John's, Newfoundland and Labrador
  - Dr. Juris Lazovskis Inc. /ID# 224817, Sydney, Nova Scotia
  - Dr. Viktoria Pavlova Medicine Professional Corporation /ID# 224536, Ancaster, Ontario
  - Drs. Rai & Sekhon Medicine Professional Corporation /ID# 224366, Brampton, Ontario
  - Dr. Sankalp V. Bhavsar Medicine Professional Corporation /ID# 223952, Burlington, Ontario
  - Paolo Pace Medicine Professional Corporation /ID# 234057, Cambridge, Ontario
  - Dr. Chrisostomos Kouroukis & Dr. Pauline Boulos MPC /ID# 223814, Dundas, Ontario
  - Arthur Karasik Medicine Professional Corporation /ID# 225276, Etobicoke, Ontario
  - Adachi Medicine Prof. Corp /ID# 223872, Hamilton, Ontario
  - St. Joseph's Healthcare /ID# 224042, Hamilton, Ontario
  - West Mountain Medical Center /ID# 222975, Hamilton, Ontario
  - Brandusa Florica Medicine Professional Corporation /ID# 222173, Mississauga, Ontario
  - Credit Valley Rheumatology /ID# 219226, Mississauga, Ontario
  - Imtiaz MS Khan Medicine Prof /ID# 225275, Mississauga, Ontario
  - Rajwinder S. Dhillon Medicine /ID# 224365, Niagara Falls, Ontario
  - Makhzoum Medicine Professional Corporation /Id# 229629, Oakville, Ontario
  - Dr. S. Gill Medicine Professional Corporation /ID# 225238, Oakville, Ontario
  - The Waterside Clinic /ID# 224205, Orillia, Ontario
  - Dr. L. Lisnevskaia Medicine Professional Corporation /ID# 225645, Oshawa, Ontario
  - Angela Montgomery Medicine Professional Corporation /ID# 231142, Ottawa, Ontario
  - Niagara Peninsula Arthritis Ct /ID# 221472, St. Catharines, Ontario
  - Dr. Sabeen Anwar Medicine Professional Corporation /ID# 224797, Windsor, Ontario
  - CIUSSS de l'est de l'Ile-de-Montreal - Hopital Maisonneuve-Rosemont /ID# 225021, Montreal, Quebec
  - Rheumatology Institute of Montreal /ID# 224045, Montreal, Quebec
  - Applied Medical Informatics Research Inc. (AMIR) /ID# 224321, Montreal, Quebec
  - Clinique de Rhumatologie de Montreal /ID# 221266, Montreal, Quebec
  - CISSSBSL -Hopital regional de Rimouski /ID# 224681, Rimouski, Quebec
  - Groupe de Recherche en Maladies Osseuses Inc /ID# 222977, Sainte-Foy, Quebec
  - CIUSSS de l'Estrie - CHUS /ID# 225404, Sherbrooke, Quebec
  - Centre de Recherche Musculo-Squelettique /ID# 224513, Trois-Rivières, Quebec
  - Dr Naik-Medical Professional Corporation-Alliance Health /ID# 221195, Saskatoon, Saskatchewan
  - Rheumatology Associates /ID# 228584, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bessette L, Chan J, Chow A, Lisnevskaia L, Richard N, Fournier PA, Liazoghli D, Girard T, Haaland D. Real-World Effectiveness of Upadacitinib for Treatment of Rheumatoid Arthritis in Canadian Patients: Interim Results from the Prospective Observational CLOSE-UP Study. Rheumatol Ther. 2024 Jun;11(3):563-582. doi: 10.1007/s40744-024-00651-8. Epub 2024 Mar 11. PMID 38467912
- See also: Clinical Study Report Synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-096#additional-resources-section